CLINICAL TRIAL: NCT01259206
Title: Increased Calcaneal Spur Incidence in Patients With Obesity and Type 2 Diabetes Mellitus
Brief Title: Plantar Faciitis and Diabetes Mellitus
Acronym: No acronym
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Gulhane School of Medicine, Department of Endocrinology and Metabolism
Other Study IDs: 11.10.2008/127
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2008-10

CONDITIONS: Diabetes Mellitus
Keywords: Calcaneal Spur, Diabetic Obese Patients
MeSH Terms: conditions — Diabetes Mellitus; Heel Spur

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- diabetic patients
- diabetic patients and healty controls: there are two groups in this study. One group is obese type 2 diabetic patiens and other group is healty controls.

SUMMARY:
Obesity is a risk factor for calcaneal spur (CS) formation which is supposed to originate from chronic plantar fasciitis. Diabetes mellitus may contribute to the risk of CS by decreased ability of tissue repair and increased reactive ossification. Thus, the investigators aimed to determine CS incidence in asymptomatic obese subjects with and without type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
OBJECTIVE-Obesity is a risk factor for calcaneal spur (CS) formation which is supposed to originate from chronic plantar fasciitis. Diabetes mellitus may contribute to the risk of CS by decreased ability of tissue repair and increased reactive ossification. Thus, the investigators aimed to determine CS incidence in asymptomatic obese subjects with and without type 2 diabetes mellitus (T2DM).

RESEARCH DESIGN AND METHODS-Ninety-three obese patients with T2DM and forty-two obese subjects without any metabolic disturbances as control were evaluated with lateral calcaneal x-ray in blinded fashion by a radiologist. All participants were informed and written consents have been obtained. Control cases were subjected to 75g glucose challenge test and glucose intolerant subjects were excluded.

RESULTS-T2DM and control groups were statistically similar in mean age (59±10.5 vs. 55±8 yrs, P=0.196, respectively) and mean body mass index (BMI)(35.1±4.3 vs. 33.1±3.3 kg/m2, P=0.073, respectively). Existence of calcaneal spur was 72% in 93 patients (77%) in T2DM group and 24 in 42 (57%) in control group. Groups were significantly different according to existence of CS (P=0.023). Mean age and mean BMI were significantly higher in diabetic patients with calcaneal spur than diabetic patients without calcaneal spur (p=0.001 and p=0.015, respectively). There was positive correlation between existence of calcaneal spur and peripheral neuropathy (p=0,043) in diabetics but no significant relation between existence of CS and glycolysed hemoglobin levels or diabetes duration (all P>0.05).

CONCLUSIONS-Clinicians should pay attention the increased incidence of CS in patients with T2DM to avoid foot complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Diabetes mellitus
* Must be obese

Exclusion Criteria:

* Previous radiotherapy to the foot,
* previous trauma to the foot (fracture, rupture of tendon),
* rheumatic or vascular diseases,
* malign diseases,
* lymphatic edema.

Ages: 49 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 93 paitents and 42 control group
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2009-02; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Increased Calcaneal Spur Incidence in Patients With Obesity and Type 2 Diabetes Mellitus | 3 months
  Calcaneal spur incidence is increased in patients with diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Aydoğan Aydoğdu, Principal Investigator — No organizational affiliation
Locations (1):
- Gulhane School of Medicine Etlik, Ankara, Turkey (Türkiye)